CLINICAL TRIAL: NCT02311257
Title: Survey on Supplement Use in Mitochondrial Disease
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: NAMDC7411
Record Dates: First submitted 2014-09-12; First posted 2014-12-08 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Mitochondrial Disease
MeSH Terms: conditions — Mitochondrial Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to learn about the use of nutritional supplements in patients with mitochondrial disease.

DETAILED DESCRIPTION:
Our goal is to better assess which nutritional supplements are prescribed to patients with mitochondrial disorders, the monitoring obtained and whether any subjective improvements are noted by the patients or their caregivers.

ELIGIBILITY:
Inclusion Criteria:

* NAMDC Clinical Registry or RDCRN Contact Registry participant
* Diagnosis of a mitochondrial disease confirmed by either electron transport chain abnormalities or molecular testing.

Exclusion Criteria:

* Lack of participation in NAMDC or RDCRN registries
* Diagnosis of mitochondrial disorder not confirmed by ETC studies or molecular diagnosis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recruited through the NAMDC Clinical Registry and RDCRN Contact Registry. Additional means of recruitment may be used to direct patients to join the NAMDC or RDCRN registries.
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Assessment of nutritional supplement use in patients with mitochondrial disease. | Up to one year after study activation.
  This cross-sectional survey will assess nutritional supplements used by patients with mitochondrial disease.

SECONDARY OUTCOMES:
Assess the attitudes of patients and parents towards use of nutritional supplements in patients with mitochondrial disease | Upt to one year after study activation.
  This cross-sectional survey will assess patients' and parents' attitudes (comfort level and perceptions of efficacy) of use of nutritional supplements in patients with mitochondrial disease.

CONTACTS AND LOCATIONS:
Overall Officials: Sumit Parikh, MD, Study Chair — The Cleveland Clinic; Amel Karaa, MD, Study Chair — Massachussetts General Hospital; Michio Hirano, MD, Study Chair — Columbia University
Locations (1):
- University of South Florida, Tampa, Florida, United States

REFERENCES:
- See also: Rare Diseases Clinical Research Network NAMDC page — http://www.rarediseasesnetwork.org/namdc/